CLINICAL TRIAL: NCT01705223
Title: Phase IIa Study of AIDS Vaccine (Combined Use of DNA Vaccine and Recombinant Vaccinia Virus Tiantan)
Brief Title: Safety and Immunogenicity Study of AIDS Vaccine (Combined Use of DNA Vaccine and Recombinant Vaccinia Virus Tiantan)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: X111012202
Record Dates: First submitted 2012-09-12; First posted 2012-10-12 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2014-10

CONDITIONS: AIDS
Keywords: prophylactic; vaccine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Vaccines, DNA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- group A (Experimental): DNA vaccine prime at week 0,4,8 and rTV boost at week 16
  Interventions: Biological: DNA vaccine; Biological: rTV boost
- group B (Experimental): DNA vaccine prime at week 0,4,8 and rTV boost at week 24
  Interventions: Biological: DNA vaccine; Biological: rTV boost
- group C (Experimental): DNA vaccine prime at week 0,4,8 and rTV boost at week 32
  Interventions: Biological: DNA vaccine; Biological: rTV boost
- group D (Experimental): DNA vaccine prime with the addition of electroporation at week 0, 4, 8 and rTV boost at week 24
  Interventions: Biological: DNA vaccine prime with the addition of electroporation; Biological: rTV boost

INTERVENTIONS:
Biological: DNA vaccine — 4mg/dose, three doses at week 0,4,8
  Arms: group A; group B; group C
Biological: DNA vaccine prime with the addition of electroporation — 4mg/dose, three doses at week 0,4,8
  Arms: group D
Biological: rTV boost — at week 16
  Arms: group A
Biological: rTV boost — at week 24
  Arms: group B; group D
Biological: rTV boost — at week 32
  Arms: group C

SUMMARY:
This trial studies the safety and immunogenicity of a HIV clade B'/C DNA vaccine followed by recombinant vaccinia virus rTV boost in HIV-uninfected healthy volunteers at low or high risk of HIV infection. In addition, the effect of different intervals of the prime-boost will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be followed for the planned duration of the study, and receive intravenous blood collection and sample storage in the 16~20 months after first vaccination;
* Understand and agree with the content of informed consent;
* Volunteers at low risk of HIV infection, or high-risk men who have sex with men (MSM）, who had have oral sex or anal sex with another man in the past 6 months ;
* Willing to be tested for HIV and syphilis;
* Before 2 weeks of the first vaccination and after 12 months of the last vaccination, willing to use an effective method of contraception with sexual partner. Female subjects are willing to undergo urine pregnancy test before each vaccination and at the follow-up visit.

Exclusion Criteria:

* Have close contact with people who are pregnant or lactating in the one month after vaccination of rTV vaccine;
* Have listed diseases or medical history:

  * Have innate or acquired immune deficiency disease or have close contact with patients suffering from the above-mentioned diseases within 1 month of rTV vaccination;
  * Need treatment affecting immunization, e.g. use corticosteroids for more than 2 weeks or use immunosuppressives, e.g. alkylating, anti-metabolite or radiotherapy, etc.; or have close contact with patients suffering from the above-mentioned diseases within 1 month of rTV vaccination;
  * Suffering from immunosuppressive diseases such as cancer, organ or stem cell transplants, non-agammaglobulinemia, etc.; or have close contact with patients suffering from the above-mentioned diseases within 1 month of rTV vaccination;
  * Past or current suffering from eczema or atopic dermatitis; currently suffering from diseases that cause skin damage such as: burns, scald, chicken pox, impetigo, shingles, psoriasis, etc.; or have close contact with patients suffering from the above-mentioned diseases within 1 month of rTV vaccination;
  * Past or current high blood pressure, heart disease, diabetes, thyroid disease, asthma, angioedema, asplenia syndrome, mental illness, epilepsy, severe anemia, leukopenia and thrombocytopenia, etc.;
  * History of syncope after vaccination or allergies;
  * Currently suffering from acute infectious diseases and febrile diseases；
* The following circumstances are:

  * Live attenuated vaccine received within 2 months or other vaccine within 2 weeks prior to enrollment;
  * Immunoglobin or blood products received within 4 months prior to enrollment;
  * Participation in another trial of a medicinal product, completed less than 30 days prior to enrollment;
  * Drug abuse, alcoholism, heavy smokers；
* The following laboratory test abnormalities, except for the results that are assessed by researchers as being no clinical significance：

  * HIV diagnostic assay positive or suspicious, HIV RNA diagnostic assay positive;
  * Anti-DNA antibody or anti-nuclear antibody positive;
  * Other laboratory test abnormalities;
* Not complying with study protocol or not obtaining informed consent because of medical, spiritual, social, occupational, and/or other reasons.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of local and general adverse events | 14-day follow-up after DNA vaccine vaccination
Occurrence and relationship to vaccination of any serious AEs (SAEs) | During the study period (Month 0-20)
Occurrence, intensity and relationship to vaccination of clinically significant abnormal haematology and biochemistry values (grade 4) | During the study period (Month 0-20)
test HIV specific T cell response by ELISPOT | 2wk, 4wk, 14wk, 24wk after rTV vaccination
test HIV specific antibody by ELISA | 2wk, 4wk, 14wk, 24wk, 48wk after rTV vaccination
Occurrence, intensity and relationship to vaccination of local and general adverse events | 28-day follow-up after rTV vaccination

SECONDARY OUTCOMES:
test HIV specific T cell response by ICS | 4wk, 8wk, 14wk, 48wk after rTV vaccination
HIV neutralizing antibody test | 4wk, 14wk, 48wk after rTV vaccination
vaccinia virus antibody test | 2wk, 4wk, 24wk after rTV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wu, M.D., Principal Investigator — Beijing YouAn Hospital; Tong Zhang, M.D., Principal Investigator — Beijing YouAn Hospital; Yiming Shao, Ph.D., Principal Investigator — NCAIDS, China CDC
Locations (1):
- Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality, China